CLINICAL TRIAL: NCT03603067
Title: A Prospective, Non-randomized, Controlled Study: To Evaluate the Psychological Status of Monophthalmic Patients Before and After Ocular Surgery
Brief Title: The Study of Psychological Status in Monophthalmic Patients With Ocular Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: SHIRB2018018
Record Dates: First submitted 2018-07-07; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Psychology, Social; Surgery
Keywords: monophthalmos; social psychology; ocular surgery
MeSH Terms: conditions — cyclopia sequence | interventions — Ophthalmologic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- monophthalmic group: The BCVA of the worse eye is less than 0.05 or CFOV is less than 5°. The better eye need to receive ocular surgery.
  Interventions: Procedure: Ocular surgery
- Normal group: The BCVA of the worse eye is more than 0.3 and CFOV is more than 10°. One of two eyes need to receive ocular surgery.
  Interventions: Procedure: Ocular surgery

INTERVENTIONS:
Procedure: Ocular surgery — Different ocular surgeries (including vitreoretinal surgery, cataract surgery, anti-glaucoma surgery etc) will be performed in one eye of the patient. In monophthalmic patient group the surgery will be performed in eye with better visual acuity.

SUMMARY:
This study is designed to evaluate the change of psychological status before and after surgery in monophthalmic patients who receive the ocular surgery in eye with better vision.

DETAILED DESCRIPTION:
Monophthalmos means the best corrected visual acuity (BCVA) of the worse eye is less than 0.05 or the central visual field (CFOV) is less than 5°. The ocular surgery of the better eye in monophthalmic patients is of high risk. On the one hand the surgical failure will result in the patient falling into permanent darkness. On the other hand the monophthalmic patient may have the same disease in both two eyes such as high axial myopia, uveitis and glaucoma, which will increase the surgical risk. There is still no consensus on whether it is necessary to take risks to perform this kind of operation. In this study we will evaluate the change of psychological status before and after surgery in monophthalmic patients who receive the ocular surgery in eye with better vision. The necessity of the ocular surgery in monophthalmic patients will be evaluated from the point of social psychology.

ELIGIBILITY:
Inclusion Criteria:

* Intention to receive ocular surgery in one of two eyes.
* Free from prior mental disorders.
* Without general disease and can tolerate the operation.
* Communication without difficulty.

Exclusion Criteria:

* With prior mental disorders.
* Can not tolerate the operation.
* Communication with difficulty.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Shanghai Aier Eye Hospital and are intended to receive ocular surgery in one of two eyes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of anxiety | Change from Baseline HAMA score at 6 months.
  Hamilton anxiety scale（HAMA）will be filled in by each patient and the final score will be recorded. The total score ranges from 0-56. A score less than 7 means no symptom of anxiety. A score between 7 to 14 means possible anxiety. A score between 14-21 means mild anxiety. A score between 21-29 means moderate anxiety. A score more than 29 means severe symptom of anxiety.
Level of depression | Change from Baseline HAMD score at 6 months.
  Hamilton depression scale (HAMD) will be filled in by each patient and the final score will be recorded. The total score ranges from 0-56. A score less than 8 means no symptom of depression. A score between 8 to 35 means mild or moderate depression. A score more than 35 means severe symptom of depression.

SECONDARY OUTCOMES:
Level of social support | Change from Baseline SSRS score at 6 months.
  Social support rating scale (SSRS) will be filled in by each patient and the final score will be recorded.

OTHER OUTCOMES:
Visual function | One day before surgery and one day, one months, three months and six months after surgery.
  BCVA and intraocular pressure (IOP) wlll be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Li, Study Director — Shanghai Aier Eye Hospital
Locations (1):
- Shanghai Aier Eye Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be partly shared in published papers.

REFERENCES:
- [Background] Hirneiss C, Neubauer AS, Herold TR, Kampik A, Hintschich C. Utility values in patients with acquired anophthalmus. Orbit. 2009;28(6):332-6. doi: 10.3109/01676830903104702. PMID 19929654